CLINICAL TRIAL: NCT00544908
Title: A Phase II Clinical Trial of Dasatinib in Patients With Metastatic Pancreatic Cancer
Brief Title: Dasatinib in Treating Patients With Stage IV Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Toxicity
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07024; P30CA033572 (NIH); CHNMC-07024; BMS-CA180-114; CDR0000570288 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2007-10-13; First posted 2007-10-16 (Estimated); Results first posted 2015-09-17 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-09

CONDITIONS: Pancreatic Cancer
Keywords: stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Dasatinib; Immunoenzyme Techniques; Immunohistochemistry

ARMS (1):
- Dasatinib (Experimental): Dasatinib 70 mg po bid (1 cycle=28 days)
  Interventions: Drug: dasatinib; Other: immunoenzyme technique; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: dasatinib
Other: immunoenzyme technique
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Dasatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well dasatinib works in treating patients with stage IV pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the 4-month progression-free survival (PFS) rate in patients with stage IV pancreatic cancer treated with dasatinib.

Secondary

* To evaluate the response rate (complete and partial response) in patients treated with this drug.
* To evaluate the median PFS and overall survival of patients treated with this drug.
* To study the toxicities and tolerability of this drug in these patients.
* To evaluate the impact of this drug on quality of life measures.
* To evaluate the impact of this drug on Src and FAK in peripheral blood mononuclear cells prior to and during treatment.
* To study the pre-treatment expression of various signaling molecules in the Src and STAT3 pathways and attempt to identify a relationship between these findings and the aggressiveness of the tumor or its response to treatment with dasatinib.

OUTLINE: This is a multicenter study.

Patients receive oral dasatinib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo tumor tissue and blood sample collection periodically for correlative and biological studies. Blood samples are analyzed for phosphorylation levels of proteins, including phospho-Src, phospho-Fak, and other relevant biomarkers, by western blotting. Tumor tissue samples are analyzed for biomarkers by immunohistochemistry.

Quality of life is assessed at baseline, after every other course during treatment, and then at 1 year after treatment using the FACT-HEP questionnaire.

After completion of study treatment, patients are followed every 2 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically* confirmed pancreatic cancer

  * Stage IV disease NOTE: *If biopsy was performed at an outside facility, the histology must be reviewed and confirmed by the Division of Pathology at the City of Hope

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Life expectancy ≥ 3 months
* Platelet count ≥ 100,000/μL
* Absolute neutrophil count ≥ 1,500/μL
* Bilirubin ≤ 1.5 mg/dL
* ALT and AST ≤ 2.5 times upper limit of normal (ULN)
* Creatinine ≤ 1.5 mg/dL and/or creatinine clearance > 60 mL/min
* PT and PTT ≤ 1.5 times ULN
* Able to swallow dasatinib whole
* No other malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix, uterus, or bladder
* No concurrent medical condition which may increase the risk of toxicity, including any of the following:

  * Pleural or pericardial effusion of any grade
  * Clinically significant coagulation or platelet function disorder (e.g., known von Willebrand's disease)
* None of the following cardiac conditions:

  * Uncontrolled angina, congestive heart failure, or myocardial infarction within the past 6 months
  * Prolonged QTc interval (i.e., QTc > 450 msec) on electrocardiogram
  * History of clinically significant ventricular arrhythmias (i.e., ventricular tachycardia, ventricular fibrillation, or Torsades de pointes)
* No hypokalemia or hypomagnesemia that cannot be corrected
* No severe infection requiring treatment
* Completely recovered from other concurrent illnesses, as deemed by the investigator
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* Recovered from prior major surgery
* No prior irradiation to the planned field
* No prior chemotherapy for pancreatic cancer
* At least 7 days since prior and no concurrent medications that may prolong the QT interval, including any of the following:

  * Quinidine
  * Procainamide
  * Disopyramide
  * Amiodarone
  * Sotalol
  * Ibutilide
  * Dofetilide
  * Erythromycin
  * Clarithromycin
  * Chlorpromazine
  * Haloperidol
  * Mesoridazine
  * Thioridazine
  * Pimozide
  * Cisapride
  * Bepridil
  * Droperidol
  * Methadone
  * Arsenic
  * Chloroquine
  * Domperidone
  * Halofantrine
  * Levomethadyl
  * Pentamidine
  * Sparfloxacin
  * Lidoflazine
* At least 7 days since prior and no concurrent potent CYP3A4 inhibitors
* At least 7 days since prior and no concurrent medications that directly and durably inhibit platelet function, including any of the following:

  * Aspirin or aspirin-containing combinations
  * Clopidogrel
  * Dipyridamole
  * Tirofiban
  * Dipyridamole
  * Epoprostenol
  * Eptifibatide
  * Cilostazol
  * Abciximab
  * Ticlopidine
  * Cilostazol
* No concurrent anticoagulants, including warfarin or heparin/low molecular weight heparin (e.g., danaparoid, dalteparin, tinzaparin, or enoxaparin)

  * Low-dose warfarin for prophylaxis to prevent catheter thrombosis or heparin for flushes of IV lines allowed
* No concurrent IV bisphosphonates during the first 8 weeks of dasatinib therapy
* No concurrent Hypericum perforatum (St. Johns wort)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-09; Primary Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Chung, MD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (2):
- United States (2):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope Medical Group, Pasadena, California

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dasatinib
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dasatinib
Number analyzed (Participants) | 7
Age, Continuous [Median (Full Range); unit: years] | 61 [41 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Rate at 4 Months
Description: Progressive disease - appearance of one or more new lesions. Unequivocal progression of existing non-target lesions. Although a clear progression of non-target lesions only is exceptional, in such circumstances, the opinion of the treating physician should prevail and the progression status should be confirmed later on by a review panel (or study chair/primary investigator).
Time Frame: Four months.
Measure: Number; unit: percentage of participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 7
percentage of participants | 0

2. Secondary Outcome: Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: After every two cycles, up to 5 years
Measure: Number; unit: percentage of participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 7
percentage of participants | 0

ADVERSE EVENTS:
Time Frame: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Description: Adverse events recorded over a period of 13 months.
Arm/Group | Dasatinib
Serious Adverse Events (participants affected / at risk) | 2/7
Other Adverse Events (participants affected / at risk) | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib (N=7)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib (N=7)
Hemoglobin decreased (Blood and lymphatic system disorders) | 5 (6)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Vitreous hemorrhage (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (2)
Gastritis (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 4 (4)
Disease progression (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 4 (5)
Flu-like symptoms (General disorders) | 1 (1)
Irritability (General disorders) | 1 (1)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (4)
Alkaline phosphatase increased (Investigations) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 4 (5)
Bilirubin increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 4 (4)
Lymphocyte count decreased (Investigations) | 2 (3)
Weight loss (Investigations) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (4)
Blood glucose increased (Metabolism and nutrition disorders) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Serum albumin decreased (Metabolism and nutrition disorders) | 2 (2)
Serum calcium decreased (Metabolism and nutrition disorders) | 2 (2)
Serum magnesium increased (Metabolism and nutrition disorders) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (2)
Bladder hemorrhage (Renal and urinary disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
Study was terminated early due to toxicity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes